CLINICAL TRIAL: NCT03288857
Title: Comparison of the Bulb Aspirator to a Nasal Oral Aspirator in the Treatment of Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Dell Children's Medical Center of Central Texas (Other)
Responsible Party: Principal Investigator, Whitney Schwarz, Principle Investigator, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-06-0086
Record Dates: First submitted 2017-09-13; First posted 2017-09-20 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Bronchiolitis; Aspirator
Keywords: Naspira; Suctioning; Nasal suction device; Children
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bulb Aspirator (No Intervention): If randomized to the bulb aspirator group, the patient will be sent home with a bulb aspirator to use for home nasal secretion management
- Nasal Oral Aspirator (NeilMed Naspira) (Experimental): If randomized to the nasal oral aspirator group, patient will be sent home with a nasal oral aspirator to use for home nasal secretion management
  Interventions: Device: NeilMed Naspira

INTERVENTIONS:
Device: NeilMed Naspira — NeilMed Naspira is a nasal-oral aspirator
  Arms: Nasal Oral Aspirator (NeilMed Naspira)

SUMMARY:
The investigators aim to compare the standard bulb aspirator with that of a nasal oral aspirator. The hypothesis is that use of a nasal oral aspirator is more effective at removing nasal secretions in the treatment of bronchiolitis as measured by a predicted 50% decrease in the rate of unscheduled bronchiolitis return visits. The primary endpoint will be the number of unscheduled bronchiolitis return visits; secondary endpoints will include measurements of oral intake, respiratory relief, parental device preference and adverse events.

DETAILED DESCRIPTION:
This study will be a single center, single blind, randomized controlled trial in the pediatric emergency department (ED) at Dell Children's Medical Center of Central Texas (DCMC). An ED discharge diagnosis of bronchiolitis will trigger patients to be randomized to receive a bulb aspirator or nasal oral aspirator for home secretion management use. Prior to dispensing the randomized aspirator, a pre-distribution questionnaire will be administered. Additionally, patients will receive a diary to complete for 3 days post ED discharge. Research personnel will call families on day 4 as a reminder to return the diary and again on day 14 to obtain a verbal post-study questionnaire. Research personnel will perform chart review on all patients looking for unscheduled patient return visits for bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

* Children >28 days of life to < 2 years of age discharged home from the DCMC ED with a diagnosis of bronchiolitis (diagnosis made per provider discretion)
* Caregiver fluent in English or Spanish

Exclusion Criteria:

* Previous enrollment
* Hospital admission
* Parental refusal to be randomized to an aspirator device (i.e., family prefers current device and does not wish to be randomized to a potentially different product)
* Current bacterial pneumonia
* Diagnosis of asthma
* Chronic lung disease
* Significant underlying cardiac disease
* Chronic neuromuscular disease

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 236 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
Unscheduled bronchiolitis return visits | 14 days
  The number of unscheduled bronchiolitis return visits (return to either ED, urgent care or PCP)

SECONDARY OUTCOMES:
Oral intake | 14 days
  Effects of device on oral intake as determined by diary and post-study questionnaire
Respiratory relief | 14 days
  Effects of device on respiratory relief as determined by diary and post-study questionnaire
Parental device preference | 14 days
  Parental device preference as determined by diary and post-study questionnaire
Adverse events | 14 days
  Description of adverse events as determined by diary and post-study questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Dell Children's Medical Center of Central Texas, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schwarz WW, Wilkinson M, Allen A. Randomized Controlled Trial Comparing the Bulb Aspirator With a Nasal-Oral Aspirator in the Treatment of Bronchiolitis. Pediatr Emerg Care. 2022 Feb 1;38(2):e529-e533. doi: 10.1097/PEC.0000000000002372. PMID 35100758